CLINICAL TRIAL: NCT07407491
Title: Comparative Efficacy Of Intraductal Antibiotic During ERCP In Acute Cholangitis: A Randomized Controlled Trial
Brief Title: Comparative Efficacy Of Intraductal Antibiotic During ERCP In Acute Cholangitis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National University of Malaysia (Other)
Responsible Party: Principal Investigator, Prof Madya Dr. Azlanudin Azman, Associate Professor, National University of Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JEP-2024-337
Record Dates: First submitted 2026-01-23; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Acute Cholangitis; Biliary Tract Infection; Biliary Obstruction; Choledocholithiasis; Malignant Biliary Stricture
Keywords: Acute Cholangitis; ERCP; Intraductal antibiotics; Biliary tract infection; Choledocholithiasis
MeSH Terms: conditions — Cholangitis; Choledocholithiasis | interventions — Gentamicins

STUDY DESIGN:
Intervention Model Description: Patients will be randomised into the intervention or control group (Intervention group will receive intraductal antibiotic Gentamicin and control group will receive intraductal distilled water in ERCP)
Who Masked: Participant, Care Provider
Masking Description: Care provider and patients are blinded from knowing the group of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gentamicin arm (Experimental): In all cases of interventional ERCP, the endoscopist will routinely administer 20cc of distilled water into the bile duct before insertion of the biliary stent or, in cases where a stent is not indicated, before withdrawal of the cannulation catheter from the bile duct to flush out remaining contrast material, sludge, or debris from the bile duct. In this study, the subjects will instead be randomized to receive either 20cc of distilled water as per usual protocol (control arm) or 20cc of intraductal antibiotic (study arm).
  Patients will receive intraductal antibiotic Gentamicin 80mg(2ml) diluted in 20cc distilled water during ERCP.
  Interventions: Drug: Gentamicin - single dose
- Distilled water arm (Active Comparator): In all cases of interventional ERCP, the endoscopist will routinely administer 20cc of distilled water into the bile duct before insertion of the biliary stent or, in cases where a stent is not indicated, before withdrawal of the cannulation catheter from the bile duct to flush out remaining contrast material, sludge, or debris from the bile duct. In this study, the subjects will instead be randomized to receive either 20cc of distilled water as per usual protocol (control arm) or 20cc of intraductal antibiotic (study arm).
  Patients will receive intraductal distilled water 20cc during ERCP.
  Interventions: Drug: Distilled water

INTERVENTIONS:
Drug: Gentamicin - single dose — Administration described in arm/group description
  Arms: Gentamicin arm
Drug: Distilled water — Administration described in arm/group description
  Arms: Distilled water arm

SUMMARY:
Does intraductal administration of antibiotics during endoscopic retrograde cholangiopancreatography (ERCP), in addition to standard systemic antibiotic therapy, improve clinical outcomes in patients with acute cholangitis compared with standard systemic antibiotic therapy alone?

DETAILED DESCRIPTION:
Acute cholangitis is a serious infection of the biliary system caused by biliary obstruction and infected bile, which may rapidly progress to sepsis if not promptly treated. Standard management includes systemic antibiotics and urgent biliary drainage, most commonly by endoscopic retrograde cholangiopancreatography (ERCP). However, biliary obstruction may impair biliary excretion of systemically administered antibiotics, resulting in subtherapeutic antibiotic concentrations within infected bile. Intraductal administration of antibiotics during ERCP may achieve higher local antimicrobial concentrations at the site of infection. This study evaluates the efficacy and safety of intraductal antibiotic administration during ERCP as an adjunct to standard systemic antibiotic therapy in patients with acute cholangitis.

ELIGIBILITY:
Inclusion Criteria:

* The patients diagnosed with mild and moderate acute cholangitis based on TG 18
* Planned for ERCP within 48 hours
* 18 years old and above

Exclusion Criteria:

* Severe acute cholangitis
* History of antibiotic hypersensitivity
* Receiving cancer chemotherapy, steroids, or immunosuppressive agents
* Concomitant infections
* Recent biliary interventions such as percutaneous transhepatic biliary drainage (PTBD) within last 3 months
* Known or suspected perforated tympanic membrane, myasthenia gravis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2024-07-09 (Actual); Primary Completion 2026-07-08 (Estimated); Study Completion 2026-07-08 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of local intraductal antibiotic administration during ERCP in patients with acute cholangitis, as assessed by resolution of clinical symptoms and improvement in inflammatory markers and liver function tests. | Evaluated at specific timepoints at admission, on the day of ERCP (pre-procedure), and daily from Day 1 to Day 3 following ERCP.
  1. Change in Inflammatory Markers: Reduction in total white cell count (WCC), expressed in ×10⁹/L, and C-reactive protein (CRP), expressed in mg/L, measured from baseline (pre-ERCP) to 24-72 hours post-ERCP.
  2. Change in Liver Function Tests: Improvement in liver function parameters including total bilirubin (µmol/L), direct bilirubin (µmol/L), alkaline phosphatase (ALP; U/L), alanine aminotransferase (ALT; U/L), aspartate aminotransferase (AST; U/L), and international normalized ratio (INR), measured from baseline (pre-ERCP) to 24-72 hours post-ERCP.
  3. Change in Vital Signs: Serial improvement in vital signs, including body temperature (°C), blood pressure (mmHg), and pulse rate (beats per minute), measured from baseline (pre-ERCP) to 72 hours following ERCP.

SECONDARY OUTCOMES:
To compare the length of hospital stay | From hospital admission through hospital discharge during the index hospitalization (up to approximately 30 days).
  Total duration of hospitalization, calculated as the number of days from the date of hospital admission to the date of hospital discharge following the index ERCP procedure.
To compare the duration of intravenous antibiotic therapy. | From initiation of intravenous antibiotic therapy after hospital admission through discontinuation of intravenous antibiotics during the index hospitalization (up to approximately 30 days).
  Criteria for intravenous to per oral switch antibiotic:
  * Able to tolerate oral therapy
  * No vomiting or diarrhea or nil by mouth
  * Clinical improvement with temperature less than 38°C, systolic blood pressure >90 mmHg, heart rate <100 beats per minute, and normal white blood cell count or a decrease of at least 2x10^9/L over the last 24 hours.
To compare the number of participants that developed a peri-procedural complication. | Evaluated at specific timepoints during the procedure until day 3 following ERCP.
  Peri-procedural complications assessed by post-ERCP monitoring, including pancreatitis, procedure-related bleeding, cardiopulmonary complications, gastrointestinal perforation, and sedation-related adverse events, recorded until day 3 following ERCP.

CONTACTS AND LOCATIONS:
Overall Officials: Azlanudin Azman, Principal Investigator — Universiti Kebangsaan Malaysia Medical Centre
Locations (1):
- Hospital Canselor Tuanku Muhriz UKM, Cheras, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Shrayteh ZM, Rahal MK, Malaeb DN. Practice of switch from intravenous to oral antibiotics. Springerplus. 2014 Dec 9;3:717. doi: 10.1186/2193-1801-3-717. eCollection 2014. PMID 25674457
- [Result] Blenkharn JI, Habib N, Mok D, John L, McPherson GA, Gibson RN, Blumgart LH, Benjamin IS. Decreased biliary excretion of piperacillin after percutaneous relief of extrahepatic obstructive jaundice. Antimicrob Agents Chemother. 1985 Dec;28(6):778-80. doi: 10.1128/AAC.28.6.778. PMID 4083861
- [Result] Buyukasik K, Toros AB, Bektas H, Ari A, Deniz MM. Diagnostic and therapeutic value of ERCP in acute cholangitis. ISRN Gastroenterol. 2013 Aug 13;2013:191729. doi: 10.1155/2013/191729. eCollection 2013. PMID 23997958
- [Result] Sood S, Winn T, Ibrahim S, Gobindram A, Arumugam AA, Razali NC, Yasmin P, Hidayu N, Sani H, Mustafa MH, Fatinah A, Devi A, Karim AA, Obaid KJ, Haron NH, Fitjerald H, Koshy M. Natural history of asymptomatic gallstones: differential behaviour in male and female subjects. Med J Malaysia. 2015 Dec;70(6):341-5. PMID 26988206
- [Result] Kimura Y, Takada T, Kawarada Y, Nimura Y, Hirata K, Sekimoto M, Yoshida M, Mayumi T, Wada K, Miura F, Yasuda H, Yamashita Y, Nagino M, Hirota M, Tanaka A, Tsuyuguchi T, Strasberg SM, Gadacz TR. Definitions, pathophysiology, and epidemiology of acute cholangitis and cholecystitis: Tokyo Guidelines. J Hepatobiliary Pancreat Surg. 2007;14(1):15-26. doi: 10.1007/s00534-006-1152-y. Epub 2007 Jan 30. PMID 17252293
- [Result] Wada K, Takada T, Kawarada Y, Nimura Y, Miura F, Yoshida M, Mayumi T, Strasberg S, Pitt HA, Gadacz TR, Buchler MW, Belghiti J, de Santibanes E, Gouma DJ, Neuhaus H, Dervenis C, Fan ST, Chen MF, Ker CG, Bornman PC, Hilvano SC, Kim SW, Liau KH, Kim MH. Diagnostic criteria and severity assessment of acute cholangitis: Tokyo Guidelines. J Hepatobiliary Pancreat Surg. 2007;14(1):52-8. doi: 10.1007/s00534-006-1156-7. Epub 2007 Jan 30. PMID 17252297
- [Result] Miura F, Okamoto K, Takada T, Strasberg SM, Asbun HJ, Pitt HA, Gomi H, Solomkin JS, Schlossberg D, Han HS, Kim MH, Hwang TL, Chen MF, Huang WS, Kiriyama S, Itoi T, Garden OJ, Liau KH, Horiguchi A, Liu KH, Su CH, Gouma DJ, Belli G, Dervenis C, Jagannath P, Chan ACW, Lau WY, Endo I, Suzuki K, Yoon YS, de Santibanes E, Gimenez ME, Jonas E, Singh H, Honda G, Asai K, Mori Y, Wada K, Higuchi R, Watanabe M, Rikiyama T, Sata N, Kano N, Umezawa A, Mukai S, Tokumura H, Hata J, Kozaka K, Iwashita Y, Hibi T, Yokoe M, Kimura T, Kitano S, Inomata M, Hirata K, Sumiyama Y, Inui K, Yamamoto M. Tokyo Guidelines 2018: initial management of acute biliary infection and flowchart for acute cholangitis. J Hepatobiliary Pancreat Sci. 2018 Jan;25(1):31-40. doi: 10.1002/jhbp.509. Epub 2018 Jan 8. PMID 28941329
- [Result] Lan Cheong Wah D, Christophi C, Muralidharan V. Acute cholangitis: current concepts. ANZ J Surg. 2017 Jul;87(7-8):554-559. doi: 10.1111/ans.13981. Epub 2017 Mar 24. PMID 28337833